CLINICAL TRIAL: NCT05862805
Title: The Role of Plasminogen Activator Inhibitor-1 (PAI-1), Tissue Plasminogen Activator (tPA), Tissue Factor Pathway Inhibitor (TFPI), and Endometrial Endothelial Cells in Uterine Hemostasis in Humans
Brief Title: PAI-1, tPA, TFPI and HEECs in Uterine Hemostasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Bannowb, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OHSU IRB 23749
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Menstrual Bleeding, Heavy
MeSH Terms: conditions — Menorrhagia | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy Menstrual Bleeding (Active Comparator): Participants with heavy menstrual bleeding will provide daily samples of menstrual blood for a single cycle and undergo a single endometrial biopsy for HEEC culture.
  Interventions: Procedure: Sample Collection and Endometrial Biopsy
- Regular Mensural Bleeding (Active Comparator): Participants with normal menstrual bleeding will provide daily samples of menstrual blood for a single cycle and undergo a single endometrial biopsy for HEEC culture.
  Interventions: Procedure: Sample Collection and Endometrial Biopsy

INTERVENTIONS:
Procedure: Sample Collection and Endometrial Biopsy — Participants will provide daily samples of menstrual blood for a single cycle and undergo a single endometrial biopsy for HEEC culture.

SUMMARY:
The purpose of the study is to learn more about the role of blood clotting factor proteins and cells in menstrual (period) bleeding. The investigators are hoping to identify differences in these proteins and cells in the menstrual blood of individuals with heavy periods compared to menstruating individuals who do not have heavy periods.

DETAILED DESCRIPTION:
The purpose of this study is to learn if human endometrial endothelial cells (HEECs) regulate human uterine hemostasis through the up and down-regulation of pro- and anti-coagulant factors in menstrual blood including PAI-1, factor XI (FXI)-PAI-1 complex, tPA, and TFPI.

This study will enroll participants with heavy menstrual bleeding (HMB) and participants without HMB. Coagulation factors will be measured in menstrual blood and mRNA for these factors will be quantified from cultured HEECS from endometrial biopsies and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Regularly menstruating participants between 18-45 years of age

Exclusion Criteria:

* Pregnancy within 3 months of enrollment
* Lactating at the time of enrollment
* Hormonal contraceptive use or use of the copper intrauterine device (IUD)
* Antifibrinolytic use
* Inherited or acquired bleeding disorder or anticoagulant use
* Known structural cause of HMB
* Inability to complete PBACs
* Unwilling to refrain from sexual intercourse for the two weeks prior to endometrial biopsy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Total number of mRNA copies from HEEC culture of tPA | Enrollment to 60 days
  The total number of mRNA copies of tPA in HEEC cultures from enrollment to 60 days.
Total number of mRNA copies from HEEC culture of PAI-1 | Enrollment to 60 days
  The total number of mRNA copies of PAI-1 in HEEC cultures from enrollment to 60 days.
Total number of mRNA copies from HEEC culture of TFPI | Enrollment to 60 days
  The total number of mRNA copies of TFPI in HEEC cultures from enrollment to 60 days.
Change in the numerical score of Pictorial Blood Loss Assessment | Enrollment to 60 days
  The change in the Pictorial Blood Loss Assessment Charts (PBACs) from baseline to 60 days. Participants will be asked to tally the number of pads and tampons, the level of saturation of menstrual blood on the pads or tampons, and the number of clots. Scores greater than 100 are considered diagnostic of heavy menstrual bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States